CLINICAL TRIAL: NCT07304154
Title: A Phase 1 Open-label, Multiregional, Multicenter, Basket Study Evaluating the Safety and Efficacy of KITE-363, an Autologous Anti-CD19/CD20 CAR T-cell Therapy in Participants With Relapsed/Refractory Autoimmune Neurologic Diseases
Brief Title: A Study Evaluating the Safety and Efficacy of KITE-363 in Relapsed/Refractory Autoimmune Neurologic Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-728-0204
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Myasthenia Gravis; Multiple Sclerosis
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Myasthenia Gravis; Multiple Sclerosis | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: KITE-363 (Dose Escalation) (Experimental): Participants with relapsing forms of multiple sclerosis (RMS), progressive forms of multiple sclerosis (PMS), myasthenia gravis (MG), and/or chronic inflammatory demyelinating polyneuropathy (CIDP) will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by infusion of KITE-363 chimeric antigen receptor (CAR) transduced autologous T cells at a single dose level, with different participants receiving sequential dose-escalation levels to find the Phase 1b recommended dose.
  Interventions: Biological: KITE-363; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1b: KITE-363 (Dose Expansion) (Experimental): Participants with RMS, PMS, MG, and/or CIDP will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed Phase 1a recommended dose of KITE-363 CAR T cells.
  Interventions: Biological: KITE-363; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: KITE-363 — A single infusion of CAR-transduced autologous T cells administered as intravenous infusion.
Drug: Fludarabine — Administered intravenously
Drug: Cyclophosphamide — Administered intravenously

SUMMARY:
This study will have two Phases: Phase 1a and Phase 1b. The goals of this clinical study are to learn more about the study drug KITE-363, by evaluating its safety, tolerability and efficacy in participants with relapsed/refractory autoimmune neurologic diseases.

The primary objectives of this study are:

* To evaluate the safety and tolerability of KITE-363 in participants with autoimmune neurologic diseases
* To determine the recommended dose for Phase 1b.
* To evaluate the preliminary efficacy of KITE-363 in participants with autoimmune neurologic diseases.

ELIGIBILITY:
Key Inclusion Criteria:

* Reproductive status-related eligibility and contraception requirements:

  * Participants must agree to use protocol-specified method(s) of contraception where applicable

Inclusion Criteria for multiple sclerosis (MS):

MS (Relapsing and progressive forms):

* Diagnosed with MS according to the 2017 revision of the McDonald diagnostic criteria

Relapsing forms of MS (relapsing-remitting multiple sclerosis (RRMS), active secondary-progressive multiple sclerosis (aSPMS)):

* Inadequate response to previous therapies is defined as evidence of breakthrough disease activity within 12 months prior to screening while on high efficacy disease-modifying therapy (DMT) OR Inadequate response to previous therapies defined as intolerance to ≥ 2 DMTs due to side effects prohibiting the chronic use of the DMT.
* Expanded Disability Status Scale (EDSS) 0 to 5.5

Progressive forms of MS (primary-progressive multiple sclerosis (PPMS) and non-active secondary-progressive multiple sclerosis (naSPMS)):

* Inadequate response to previous therapies is defined as evidence of disease progression within 12 months prior to screening despite standard of care therapy for naSPMS or despite ocrelizumab, where available, for PPMS
* Absence of clinical relapses for at least 24 months
* No evidence of Gadolinium enhancing (GadE+) on magnetic resonance imaging (MRI) brain at screening or baseline
* EDSS of 3 to 6.5 who are ambulatory

Inclusion Criteria for myasthenia gravis (MG):

* Documentation of autoantibodies against acetylcholine receptor (AChR), muscle-specific kinase (MuSK), or low-density lipoprotein receptor-related protein 4 (LRP4)
* Diagnosis of MG with generalized weakness meeting criteria as defined by the Myasthenia Gravis Foundation of American (MGFA) classification of II- IV at screening
* Myasthenia Gravis Activities of Daily Living (MG-ADL) score ≥ 6 (> 50% of the total score due to non-ocular symptoms)
* Quantitative Myasthenia Gravis (QMG) score ≥ 10
* Inadequate response to previous therapies while taking at least 2 classes of immunosuppressants (ie, steroids, azathioprine (AZA), mycophenolate mofetil (MMF), intravenous immunoglobulin (IVIg), biologics (eg, rituximab, anti-neonatal fragment crystallizable (Fc) receptor (FcRN) class, and anti-complement class))
* Thymectomy allowed if completed ≥ 12 months prior to screening

Inclusion Criteria for chronic inflammatory demyelinating polyneuropathy (CIDP):

* Probable or definite CIDP as defined by the 2010 European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) criteria, relapsing or progressive forms
* CIDP Disease Activity Status (CDAS) score ≥ 3 at screening
* Inflammatory neuropathy cause and treatment (INCAT) score ≥ 3
* Inadequate response to previous therapies despite standard of care therapy (ie, steroids, IVIg, subcutaneous immunoglobulin (SCIg), plasmapheresis exchange (PLEX), rituximab, or anti FcRN) OR Unable to tolerate standard of care due to side effects with ongoing disease activity
* Except for nodal/paranodal CIDP, historical documentation of objective improvement in the past 24 months while on IVIg, SCIg, PLEX, or anti-FcRN OR Historical documentation of objective disease worsening in the past 24 months when IVIg, SCIg, PLEX, or anti-FcRN has been reduced or interrupted

Key Exclusion Criteria:

* History or presence of central nervous system (CNS) or peripheral nervous system disorders before enrollment that may impact cognition, strength, or cause weakness
* History of autologous or allogeneic stem cell transplant and/or organ transplant

Exclusion Criteria for MS:

* Cohort 1 or 2; inability to complete 9-hole Peg Test (9-HPT) in < 240 seconds and Timed 25 foot Walk (T25FW) < 150 seconds
* History of hypersensitivity to parenteral administration of gadolinium-based contrast agents
* Any renal condition that would preclude the administration of gadolinium (for the relapsing forms of MS and progressive forms of MS)
* Any contraindication to lumbar puncture (LP) (for the relapsing forms of MS and progressive forms of MS)

Exclusion Criteria for MG:

* Current myasthenic crisis not effectively controlled within 2 weeks before enrollment
* Thymectomy performed within 12 months of baseline

Exclusion Criteria for CIDP:

* Pure sensory CIDP and focal CIDP
* Polyneuropathy of other causes

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Percentage of Participants Experiencing Treatment-emergent Adverse Event (TEAEs) | Up to 2 years
Phase 1a: Percentage of Participants Experiencing Dose-limiting Toxicities (DLTs) After the Infusion of KITE-363 | Up to 28 days
Phase 1b: (All Cohorts) Percentage of Participants Experiencing TEAEs | Up to 2 years
Phase 1b: Relapsing Forms of MS (RRMS) and (aSPMS): Number of New T1 Gadolinium Enhancing (GadE+) Lesions on Magnetic Resonance Imaging (MRI) at Week 12 | Week 12
  This will be reported in participants with relapsing forms of Multiple Sclerosis MS (RRMS) and (aSPMS).
Phase 1b: Relapsing Forms of MS (RRMS and aSPMS): Number of New and/or Enlarging T2 Lesions on MRI at Week 12 | Week 12
Phase 1b: Progressive Forms of MS (PPMS) and (naSPMS): Time to Onset of Confirmed Disability Progression Over 12 Weeks (CDP-12) | Up to 2 years
Phase 1b: Myasthenia Gravis (MG): Proportion of Participants of MG Activities of Daily Living (MG-ADL) Responders | Up to Week 24
  The MG-ADL is a scale to measure the functional impact of MG on daily activities. The total score ranges from 0 to 24, with higher scores indicating greater disability and disease burden.
Phase 1b: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP): Proportion of Participants with Confirmed Evidence of Clinical Improvement at Week 24 | Week 24
  Clinical improvement will be analyzed using inflammatory neuropathy cause and treatment (INCAT) scale. The INCAT score is a clinician administered tool used to assess functional disability in participants with CIDP. The total scores range from 0 to 10, higher scores indicating greater disability and lower score would indicate clinical improvement.

SECONDARY OUTCOMES:
Relapsing forms of MS (RRMS and aSPMS): Annual Relapse Rate | Up to 2 years
  Proportion of participants with annual relapse.
Relapsing Forms of MS (RRMS and aSPMS): Proportion of Participants With CDP-12 | Up to 2 years
Relapsing Forms of MS (RRMS and aSPMS): Proportion of Participants With CDP-24 | Up to 2 years
Relapsing Forms of MS (RRMS and aSPMS): Time to Onset of CDP-12 | Up to 2 years
Relapsing Forms of MS (RRMS and aSPMS): Time to Onset of CDP-24 | Up to 2 years
Progressive forms of MS (PPMS and naSPMS): Proportion of Participants with No Evidence of Disease Activity (NEDA) | Up to 2 years
Relapsing Forms of MS (RRMS and aSPMS): Change From Baseline in Expanded Disability Status Scale (EDSS) Score Over Time | Up to 2 years
  EDSS is scale used to measure disability and disease progression in participants with MS. It ranges from 0 (normal neurological exam) to 10 (death due to MS) in 0.5-point increments.
Relapsing Forms of MS (RRMS and aSPMS): Change From Baseline in Timed 25-foot Walk (T25FW) Score Over Time | Up to 2 years
  The T25FW is a performance-based measure used in people with MS to assess walking speed and mobility. Lower times indicate better walking ability, while longer times reflect greater impairment.
Relapsing Forms of MS (RRMS and aSPMS): Change From Baseline in 9-hole Peg Test Dominant/Non-dominant (9-HPT D/ND) Score Over Time | Up to 2 years
  The 9-HPT assesses hand dexterity and fine motor function by timing how long it takes a participant to place and remove nine pegs from a board. Faster times indicate better function, while slower times reflect greater disability.
Relapsing Forms of MS (RRMS and aSPMS): Change From Baseline in Symbol Digit Modalities Test (SDMT) Score Over Time | Up to 2 years
  SDMT is a performance-based cognitive assessment to measure information processing speed. The score is the number of correct responses completed in the time limit, with higher scores indicating better cognitive processing speed.
Progressive Forms of MS (PPMS and naSPMS): Proportion of Participants with CDP-12 | Up to 2 years
Progressive Forms of MS (PPMS and naSPMS): Proportion of Participants with CDP-24 | Up to 2 years
Progressive forms of MS (PPMS and naSPMS): Time to Onset of CDP-24 | Up to 2 years
Progressive forms of MS (PPMS and naSPMS): Number of new and Enlarging T2 Lesions on MRI | Up to 2 years
Relapsing forms of MS (RRMS and aSPMS): Percentage of Participants With NEDA | Up to 2 years
Progressive forms of MS (PPMS and naSPMS): Change From Baseline in EDSS Over Time | Up to 2 years
  EDSS is scale used to measure disability and disease progression in participants with MS. It ranges from 0 (normal neurological exam) to 10 (death due to MS) in 0.5-point increments.
Progressive forms of MS (PPMS and naSPMS): Change From Baseline in T25FW Over Time | Up to 2 years
  The T25FW is a performance-based measure used in people with MS to assess walking speed and mobility. Lower times indicate better walking ability, while longer times reflect greater impairment.
Progressive forms of MS (PPMS and naSPMS): Change From Baseline in 9-HPT D/ND Over Time | Up to 2 years
  The 9-HPT assesses hand dexterity and fine motor function by timing how long it takes a participant to place and remove nine pegs from a board. Faster times indicate better function, while slower times reflect greater disability.
Progressive forms of MS (PPMS and naSPMS): Change From Baseline in SDMT Over Time | Up to 2 years
  SDMT is a performance-based cognitive assessment to measure information processing speed. The score is the number of correct responses completed in the time limit, with higher scores indicating better cognitive processing speed.
MG: Proportion of Participants With at Least a 2-Point or 5 Point Improvement in MG-ADL Score up to Week 24 | Up to 24 weeks
  The MG-ADL is a scale to measure the functional impact of MG on daily activities. The total score ranges from 0 to 24, with higher scores indicating greater disability and disease burden.
MG: Change From Baseline in MG-ADL Score at Week 24 | Baseline, Week 24
  The MG-ADL is a scale to measure the functional impact of MG on daily activities. The total score ranges from 0 to 24, with higher scores indicating greater disability and disease burden.
MG: Proportion of Participants With Minimal Symptom Expression (MG-ADL Score of 0 or 1 Point) | Up to 2 years
  The MG-ADL is a scale to measure the functional impact of MG on daily activities. The total score ranges from 0 to 24, with higher scores indicating greater disability and disease burden.
MG: Proportion of Participants With at Least a 3-point or 5-point Improvement in Medical Research Council (QMG) Score up to Week 24 | Baseline, Week 24
  The QMG test is a standardized quantitative strength scoring system developed specifically for MG. The total QMG score is the sum of the scores for 13 items, with a possible maximum score of 39. A higher score indicates more severe disease involvement, while a lower score suggests less functional impairment.
MG: Change From Baseline in QMG Score to Week 24 | Baseline, Week 24
  The QMG test is a standardized quantitative strength scoring system developed specifically for MG. The total QMG score is the sum of the scores for 13 items, with a possible maximum score of 39. A higher score indicates more severe disease involvement, while a lower score suggests less functional impairment.
MG: Proportion of Participants With at Least a 3-Point Improvement in MG-C Score up to Week 24 | Baseline, Up to 24 weeks
  MG-C scale is a tool that measures disease severity in MG. The total score ranges from 0 to 50, with higher scores indicating greater impairment.
Change From Baseline in MG-C Scale Score at Week 24 | Baseline, Week 24
  MG-C scale is a tool that measures disease severity in MG. The total score ranges from 0 to 50, with higher scores indicating greater impairment.
MG: Number of Participants With Changes in Myasthenia Gravis Foundation of American Post-Intervention Status (MGFA-PIS), Including Minimal Manifestation, Complete Stable Remission, Pharmacologic Remission | Up to 2 years
  The MGFA-PIS is a standardized classification system which categorizes outcomes into distinct states such as complete stable remission (CSR), pharmacologic remission (PR), minimal manifestations (MM), improved, unchanged, worse, and exacerbation. CSR indicates no symptoms or signs for at least one year without therapy, while MM reflects minimal weakness without functional limitation.
CIDP: Time to First Adjusted INCAT Deterioration | Up to 2 years
  INCAT is a clinician-administered tool used to assess functional disability in participants with CIDP. The total score ranges from 0 to 10, where higher scores indicate greater disability and lower score would indicate clinical improvement.
CIDP: Proportion of Participants With Confirmed Evidence of Clinical Improvement | Week 48
  Clinical improvement will be analyzed using INCAT scale. The INCAT score is a clinician administered tool used to assess functional disability in participants with CIDP. The total scores range from 0 to 10, higher scores indicating greater disability and lower score would indicate improvement.
CIDP: Proportion of Participants With Evidence of Clinical Improvement | Up to week 48
  Clinical improvement will be analyzed using inflammatory Rasch-built overall disability scale (I-RODS) scale. I-RODS is a scale that assesses activity and participation limitations in people with CIDP. The score ranges from 0 to 48, with higher scores indicating better functional ability.
CIDP: Time to Disease Progression by I-RODS | Baseline, Up to 48 Weeks
  I-RODS is a scale that assesses activity and participation limitations in people with CIDP. The score ranges from 0 to 48, with higher scores indicating better functional ability.
CIDP: Change From Baseline Over Time in 24-Item I-RODS Score | Up to 2 years
  I-RODS is a scale that assesses activity and participation limitations in people with CIDP. The score ranges from 0 to 48, with higher scores indicating better functional ability.
CIDP: Change From Baseline Over Time in Medical Research Council (MRC) Sum Score | Up to 2 years
  MRC Sum Score is a measure to assess muscle strength for people with CIDP. The score ranges from 0 to 60. Higher scores indicate better muscle strength, while lower scores reflect greater weakness.
CIDP: Change From Baseline Over Time in Adjusted INCAT Score | Up to 2 years
  INCAT is a tool used to assess functional disability in participants with CIDP. The total score ranges from 0 to 10, where higher scores indicate greater disability.
CIDP: Change From Baseline Over Time in Timed Up and Go (TUG) Score | Up to 2 years
  TUG test is a measure of mobility, balance, and fall risk. The score is recorded in seconds; shorter times indicate better mobility, while longer times suggest impaired balance or gait.
CIDP: Change From Baseline Over Time in Mean grip strength assessed by Martin Vigorimeter | Up to 2 years
  Mean Grip Strength is a quantitative measure of hand and forearm muscle strength. Higher values indicate better muscle strength, while lower values reflect weakness or functional impairment.
Levels of T-cells in Blood | Up to 2 years
Pharmacokinetics: Levels of Chimeric Antigen Receptor (CAR) T-cells in Blood | Up to 2 years
Pharmacodynamics Parameters: Levels of B cells in Blood | Up to 2 years
Pharmacodynamics Parameters: Levels of Disease-Specific Biomarkers and Autoantibodies in Blood | Up to 2 years
Pharmacodynamics Parameters: Levels of Cytokines and Chemokines in Blood | Up to 2 years
  A panel of inflammatory, immuno-modulatory and effector molecules, including cytokines and chemokines, will be measured as units of concentration in serum (e.g. pg/ml) using ligand-based immunoassays such as MSD, Ella and O-link.
Proportion of Participants With of Antibodies Against the KITE-363 CAR T cells in Blood | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07304154